CLINICAL TRIAL: NCT00461903
Title: A Prospective, Randomized, Double-blind Placebo-controlled Study to Determine the Efficacy of 8 mg/Day Oral Perindopril to Prevent the Recurrence of Atrial Fibrillation in Patients With Essential Hypertension
Brief Title: Efficacy of Perindopril to Prevent Recurrence of Atrial Fibrillation in Patients With Essential Hypertension
Acronym: CTAF-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IC4-9490-123-CAN
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Essential Hypertension; Atrial Fibrillation
Keywords: essential hypertension; symptomatic paroxysmal or persistent atrial fibrillation
MeSH Terms: conditions — Essential Hypertension; Atrial Fibrillation | interventions — Perindopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (for perindopril) (Placebo Comparator): Sugar pill manufactued to mimic perindopril
  Interventions: Drug: Perindopril
- Perindopril (Active Comparator): Perindopril (coversyl) 4 mg tablets
  Interventions: Drug: Perindopril

INTERVENTIONS:
Drug: Perindopril — Perindopril 4 mg or matching placebo , 1 tablet administrated once daily for the first 2 weeks. If tolarable, dosage increased to 8mg/day until the end of the study (
  Other Names: Coversyl

SUMMARY:
The purpose of this 7- to 13-month study is to determine the efficacy of 8 mg/day oral perindopril to prevent the recurrence of atrial fibrillation (AF) in patients with essential hypertension.

DETAILED DESCRIPTION:
Hypertension affects approximately 50 million individuals in the United States and approximately 1 billion individuals worldwide. As the population ages, the prevalence of hypertension is expected to increase even further unless broad and effective preventive measures are implemented. Recent data from the Framingham Heart Study suggest that individuals who are normotensive at 55 years of age have a 90% lifetime risk for developing hypertension. The relationship between blood pressure (BP) and risk of cardiovascular disease (CVD) events is continuous, consistent, and independent of other risk factors. The higher the BP, the greater is the chance of myocardial infarction, heart failure (HF), stroke, and kidney disease.

Atrial fibrillation (AF) is also a major health problem and has been described as one of two emerging cardiovascular epidemics at the turn of the century. It is the most frequent cardiac arrhythmia, affecting 5% of individuals aged > 65 years, and it is associated with an increased risk of stroke and a doubling of all-cause mortality. The loss of effective atrial contraction may result in impaired cardiac performance, reduced exercise tolerance and congestive heart failure. In addition, patients with atrial fibrillation often have disabling palpitations.

Perindopril (Coversyl) is an angiotensin-converting enzyme (ACE) inhibitor with demonstrated efficacy in controlling hypertension. There are several lines of evidence suggesting that ACE inhibition may reduce the incidence of new-onset AF as well as AF recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be age 18 years or older.
* Patients may be either male or female without childbearing potential (or with adequate contraception).
* Patients must have a current diagnosis of essential hypertension with systolic blood pressure (SBP) ≤ 160 mmHg and diastolic blood pressure (DBP) ≤ 100 mmHg at the time of inclusion visit AND
* Patients must have had at least one episode of symptomatic paroxysmal or persistent atrial fibrillation within the preceding six months:

  * With an indication for cardioversion in the case of persistent AF
  * With electrocardiogram (ECG) documentation of AF
  * With duration of an AF episode of at least 10 minutes

Exclusion Criteria:

* Unlikely to co-operate in the study
* Pregnancy, breastfeeding, or possibility of becoming pregnant during the study (patients must have adequate contraception as determined by the investigator).
* Alcoholism or drug abuse
* Participation in another study at the same time or within 30 days of randomisation.
* Left ventricular systolic dysfunction with an ejection fraction of 45% or less
* Myocardial infarction within the past month prior to the selection visit
* Cardiac or thoracic surgery within the past 3 months or likely to be performed during the trial
* Chronic AF (continuously present for > 6 months)
* AF secondary to an acute reversible condition (e.g. post-operative atrial fibrillation, hyperthyroidism)
* Currently requiring class I or class III anti-arrhythmic drug therapy (for atrial fibrillation or any other arrhythmia)
* Any medical condition that makes the patient an unsuitable candidate in the investigator's opinion
* Any medical condition requiring ACE inhibitor or angiotensin-receptor blocker therapy (e.g. diabetes, known proteinuria of more than 300 mg per day)
* Renal insufficiency with serum creatinine of 180 μmol/L or greater
* Known bilateral renal artery stenosis
* Serum potassium of 5.0 mmol/L or greater on recent laboratory exam
* Positive pregnancy test (beta human chorionic gonadotropin [HCG] performed in women of childbearing potential)
* Known intolerance to ACE inhibitor
* Impossibility to discontinue certain treatments at selection visit
* Known contraindication(s) to perindopril
* Severe known liver disease including cirrhosis, biliary obstruction or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevation more than 3 times the upper limit of normal
* Use of ACE inhibitor or angiotensin-receptor blocker in the 3 months before the inclusion visit
* Severely uncontrolled hypertension with SBP > 160 mmHg or DBP > 100 mmHg at the inclusion visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2007-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be time to first sustained recurrence of AF. | 12 months follow-up
  1 month treatment adjustment 3 months of endpoint follow-up - M4 6 months of endpoint follow-up - M7 12 months of endpoint follow-up - M13

SECONDARY OUTCOMES:
Secondary efficacy endpoints will be the proportion of patients without AF throughout the 6 months of follow-up, number of documented relapses of AF, and health care resource utilization (including hospitalisations for AF and cardioversions). | 6 months follow-up
  Secondary efficacy endpoints will be the proportion of patients without AF throughout the 6 months of follow-up,number of documented relapses of AF, and health care resources utilization (including hospitalisations for AF and cardioversion)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Talajic, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Result] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255